CLINICAL TRIAL: NCT03227926
Title: A Phase II Trial of Rechallenge With Panitumumab Driven by RAS Clonal-mediated Dynamic of Resistance
Brief Title: Rechallenge With Panitumumab Driven by RAS Dynamic of Resistance
Acronym: CHRONOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 013-IRCC-10IIS-16; 2016-002597-12 (EudraCT Number)
Record Dates: First submitted 2017-07-18; First posted 2017-07-24 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
Keywords: RAS; Panitumumab; EGFR; Clonal evolution
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Intervention Model Description: Patiens will be first enrolled in a Molecular Screening (MS) Phase to determine the "molecular eligibility" of the patients for third line panitumumab re-challenge. During MS phase, patients will be liquid biopsied (LB) at different check-points (BML which is optional, Basal Mutational Load and RML which is mandatory, Rechallenge Mutational Load) and their ctDNA tested by ddPCR to monitor the presence of RAS and EGFR ECD altered clones. Patients with no RAS and EGFR ECD mutations in the RML will be declared "molecularly eligible" for the Trial Phase.
  Patients resulting "molecularly eligible" at the RML checkpoint, upon Informed Consent signature and having satisfied all other eligibility criteria, will be treated in the Trial Phase with panitumumab monotherapy at standard dose until documented radiological progression or unacceptable toxicity or any other reason (See Section 9.2.3) whichever comes first.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening Phase (Experimental): Patiens will be first enrolled in a Molecular Screening (MS) Phase to determine the "molecular eligibility" of the patients for third line panitumumab re-challenge. During MS phase, patients will be liquid biopsied (LB) at different check-points (BML which is optional, Basal Mutational Load and RML which is mandatory, Rechallenge Mutational Load) and their ctDNA tested by ddPCR to monitor the presence of RAS and EGFR ECD altered clones. Patients with no RAS and EGFR ECD mutations in the RML will be declared "molecularly eligible" for the Trial Phase.
  Interventions: Diagnostic Test: Molecular Screening
- Trial Phase (Experimental): Patients resulting "molecularly eligible" at the RML (Rechallenge Mutational Load) checkpoint, upon Informed Consent signature and having satisfied all other eligibility criteria, will be treated with panitumumab monotherapy at standard dose until documented radiological progression or unacceptable toxicity or any other reason whichever comes first.
  Interventions: Drug: Panitumumab 20 MG/ML Intravenous Solution [VECTIBIX]

INTERVENTIONS:
Drug: Panitumumab 20 MG/ML Intravenous Solution [VECTIBIX] — Panitumumab 6 mg/kg in 100 cc 0.9% NaCl solution on Day 1 every two weeks by IV administration over 1 hour.
  Other Names: VECTIBIX
  Arms: Trial Phase
Diagnostic Test: Molecular Screening — Patients without plasmatic evidence of potentially resistant clones harbouring RAS or EGFR-ectodomain mutations in the RML liquid biopsy, will be molecular eligible for the trial phase
  Other Names: RML Liquid Biopsies analysis
  Arms: Screening Phase

SUMMARY:
This is a hypothesis driven, open label, single-arm, multiple centers, Phase II trial. The trial has been designed to prove or disprove whether a rechallenge with panitumumab can achieve an objective response rate (ORR= CR+PR) of 30% or more in a population of RAS wild type mCRC patients selected on the basis of RAS extended clonal evolution in their plasma.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer in the world and the second leading cause of cancer death in the United States and the European Union. In the last decade, substantial advances in the treatment of the metastatic disease (mCRC) have more than doubled overall survival (OS) from 12 months to 30 months due to the refinement of fluoropirimidine-based chemotherapy and the introduction of antiangiogenics and targeted therapies.

Pharmacologic blockade of the epithelial growth factor receptor (EGFR) with specific monoclonal antibodies, namely, cetuximab and panitumumab, represents the mainstay of tumour targeted therapy for mCRC in patients with tumors not harboring extended RAS pathway mutations (KRAS, NRAS, or BRAF). Such alterations, which constitutively activate typical EGFR downstream transducers, have been shown to trigger substitute survival pathways that bypass therapeutic blockade of EGFR signalling, thus abating the efficacy of anti-EGFR antibodies ("primary resistance"). Even when response to anti-EGFR therapy occurs in the context of appropriate molecular selection, acquired ("secondary") resistance inevitably arises in all cases. Our group has extensively studied this phenomenon and has shown that extended-RAS alterations are the principal culprit of anti EGFR acquired resistance, and that altered RAS clones decay upon anti-EGFR treatment withdrawal, while tumor cells regain sensitivity to anti EGFR treatment. We have also documented that ctDNA profiles of individuals who benefit from multiple challenges with anti-EGFR antibodies, exhibit pulsatile levels of mutant KRAS. Collectively, these results indicate that the CRC genome adapts dynamically to intermittent anti-EGFR drug schedules, and provide a molecular explanation for the efficacy of re-challenge therapies based on EGFR blockade. Our results also give experimental support to the empirical-based clinical benefit observed, following cetuximab or panitumumab rechallenge in two small series of originally KRAS exon 2 wild type mCRC patients.

We propose to assess the efficacy and safety of re-challenging with panitumumab RAS-extend wild type mCRC patients with ctDNA-confirmed secondary resistance to anti EGFR treatment, after progression on second or further lines chemotherapy. As proof-of-concept, patients will be blood monitored throughout their therapeutic itinerary for the presence of extended-RAS alterations and EGFR-ectodomain mutations by ctDNA determination (liquid biopsy). We also include in our ddPCR panel 7 different EGFR extracellular domain (ECD) mutations as they occur in 15-20% of patients who acquired resistance to anti-EGFR drugs.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed diagnosis of metastatic colorectal cancer;
2. Age ≥ 18 years;
3. Written informed consent;
4. Documented WT RAS exons 2, 3 and 4 (KRas and NRas) and WT BRAF V600E for anti-EGFR treatment.
5. Complete or partial response to anti EGFR antibodies in any line either received as monotherapy or in combination with chemotherapy;
6. Imaging documented progression while on therapy with a therapeutic regimen including anti-EGFR mAb;
7. Imaging documented progression at the last treatment regimen that must be anti-EGFR free;
8. Patient must be RAS and EGFR ectodomain wild type in a liquid biopsy performed no longer that 4 weeks after progression to the last anti-EGFR free treatment
9. FFPE sample used for eligibility to anti-EGFR prescription (see criteria 4) must be available for custom gene panel profiling (as described in appendix B). Otherwise if sample is not available, center must have already perfomed a genotyping on this tissue sample according to appendix B.
10. ECOG performance status ≤ 2;
11. At least one measurable tumor lesion as per RECIST v1.1. Lesions in previously irradiated areas or those that have received other loco-regional therapies (i.e. percutaneous ablation) should not be considered measurable unless there is clear documented evidence of progression of the lesion since therapy. Imaging must be performed maximum within 28 days prior to registration;
12. Normal organ functions;
13. Negative serum pregnancy test within 1 week prior to the first study dose in all women of childbearing potential;
14. Subjects and their partners must be willing to avoid pregnancy during the trial. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception;
15. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Exclusion Criteria

1. History of severe infusion reactions to monoclonal antibodies cetuximab or panitumumab;
2. Symptomatic or untreated leptomeningeal disease and symptomatic brain metastasis;
3. Clinically significant cardiac disease including:

   1. congestive heart failure requiring treatment (NYHA grade ≥ 2), Left ventricular ejection fraction (LVEF) < 45% as determined by Multigated acquisition (MUGA) scan or echocardiogram;
   2. history or presence of clinically significant ventricular arrhythmias or atrial fibrillation;
   3. clinically significant resting bradycardia;
   4. unstable angina pectoris ≤ 3 months prior to starting study drug;
   5. acute myocardial infarction ≤ 3 months prior to starting study drug;
   6. QTcF > 480 msec;
4. History of thromboembolic or cerebrovascular events within the last 6 months, including transient ischemic attack, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism;
5. Patients with interstitial pneumonitis or pulmonary fibrosis;
6. Abnormal organ or bone marrow functions defined as:

   1. Absolute neutrophil count < 1.5 x 10/L;
   2. hemoglobin < 9 g/dL;
   3. alkaline phosphatase > 2.5 x upper normal limit (ULN), if liver metastases > 5 x ULN;
   4. aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) > 2.5 x ULN, if liver metastases > 5 x ULN;
   5. bilirubin > 1.5 x ULN, if liver metastases > 2 x ULN;
   6. serum creatinine > 1.5 x ULN and/or creatinine clearance ≤ 50 mL/min calculated according to Cockroft-Gault;
   7. Patients with platelet count <100 x 10^9/L
7. Previous or concurrent second malignancy. Exceptions: adequately treated basal cell or squamous cell skin cancer; in situ carcinoma of the cervix, treated curatively and without evidence of recurrence for at least 3 years prior to study entry; or other solid tumor treated curatively and without evidence of recurrence for at least 3 years prior to study entry.
8. Patients with positive serology for HIV, HBV, HCV.
9. Patients with a history of severe or life threatening hypersensitivity to the active substance or to any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) to panitumumab according to RECIST v1.1. | Tumor assessments every 8 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Main objective of the study is the evaluation of objective response rate according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression Free Survival | every 2 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  PFS is defined as the time from first treatment to the time of disease progression
Overall Survival | every 2 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  OS is defined as the length of time from the start of treatment to death from any cause
Toxicity according to CTCAE version 4.03. | every 2 weeks from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Toxicity will be assessed using the Common Toxicity Criteria for Adverse Events version 4.03 (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Siena, MD, Study Chair — Grande Ospedale Metropolitano Niguarda - Milano; Alberto Bardelli, MD, Study Chair — Fondazione del Piemonte per l'Oncologia; Silvia Marsoni, MD, Study Chair — Fondazione del Piemonte per l'Oncologia
Locations (4):
- Italy (4):
  - Istituto Nazionale Tumori - IRCCS, Milan, Via Giacomo Venezian, 1
  - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Oncologico Veneto - IRCCS, Padua

REFERENCES:
- [Derived] Ciardiello D, Martinelli E, Troiani T, Mauri G, Rossini D, Martini G, Napolitano S, Famiglietti V, Del Tufo S, Masi G, Santini D, Avallone A, Pietrantonio F, Lonardi S, Di Maio M, Zampino MG, Fazio N, Bardelli A, Siena S, Cremolini C, Sartore-Bianchi A, Ciardiello F. Anti-EGFR Rechallenge in Patients With Refractory ctDNA RAS/BRAF wt Metastatic Colorectal Cancer: A Nonrandomized Controlled Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245635. doi: 10.1001/jamanetworkopen.2024.5635. PMID 38592721
- [Derived] Sartore-Bianchi A, Pietrantonio F, Lonardi S, Mussolin B, Rua F, Crisafulli G, Bartolini A, Fenocchio E, Amatu A, Manca P, Bergamo F, Tosi F, Mauri G, Ambrosini M, Daniel F, Torri V, Vanzulli A, Regge D, Cappello G, Marchio C, Berrino E, Sapino A, Marsoni S, Siena S, Bardelli A. Circulating tumor DNA to guide rechallenge with panitumumab in metastatic colorectal cancer: the phase 2 CHRONOS trial. Nat Med. 2022 Aug;28(8):1612-1618. doi: 10.1038/s41591-022-01886-0. Epub 2022 Aug 1. PMID 35915157